CLINICAL TRIAL: NCT07040878
Title: Antigravity Treadmill Rehabilitation After Lower Limb Arthroplasty in Older Adults
Brief Title: Antigravity Treadmill After Joint Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Collaborators: Wroclaw Medical University (Other); Jan Dlugosz University in Czestochowa (Other)
Responsible Party: Principal Investigator, Błażej Cieślik, Professor, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KE-U/74/2025
Record Dates: First submitted 2025-06-17; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Arthropathy; Osteoarthritis
Keywords: arthroplasty; balance; fall risk; gait rehabilitation; psychological outcomes
MeSH Terms: conditions — Joint Diseases; Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Antigravity Treadmill Training Group (Experimental): Conventional orthopedic rehabilitation supplemented by antigravity yreadmill training
  Interventions: Behavioral: Antigravity Treadmill Training; Behavioral: Conventional rehabilitation
- Body Weight-Supported Treadmill Training (Active Comparator): Conventional orthopedic rehabilitation supplemented by body weight-supported treadmill training
  Interventions: Behavioral: Body Weight-Supported Treadmill Training; Behavioral: Conventional rehabilitation
- Control Group (Active Comparator): Conventional orthopedic rehabilitation
  Interventions: Behavioral: Conventional rehabilitation

INTERVENTIONS:
Behavioral: Antigravity Treadmill Training — Antigravity treadmill training uses air pressure to reduce effective body weight during walking, minimizing joint load while preserving gait mechanics. The 6-week intervention includes five sessions per week within a 120-minute daily kinesitherapy program. Treadmill speed is individualized at baseline and increased by 0.5 km/h every two weeks. Unloading is progressively reduced: 60% support in weeks 1-2, 40% in weeks 3-4, and 20% in weeks 5-6, allowing gradual adaptation to full weight-bearing.
  Arms: Antigravity Treadmill Training Group
Behavioral: Body Weight-Supported Treadmill Training — Body weight-supported treadmill training uses a harness-based system to partially offload body weight, promoting safe ambulation and gait normalization in early postoperative rehabilitation. The 6-week intervention includes five sessions per week within the 120-minute daily kinesitherapy program. Treadmill speed is individualized at baseline and increased by 0.5 km/h every two weeks, depending on tolerance. The unloading level remains constant and is individually adjusted to ensure safety.
  Arms: Body Weight-Supported Treadmill Training
Behavioral: Conventional rehabilitation — Conventional rehabilitation follows standard postoperative protocols after hip or knee arthroplasty. The 6-week program includes five weekly sessions. Gait training is conducted in hospital corridors under physiotherapist supervision, using assistive devices as needed (crutches, walkers). Daily therapy includes 120 minutes of kinesiotherapy (general exercises and gait training), 30 minutes of ergotherapy to improve functional independence, and three individualized physical therapy procedures (laser therapy, magnetic therapy, or electrotherapy) tailored to patient needs.

SUMMARY:
The study aims to evaluate the efficacy of antigravity treadmill training and body weight-supported treadmill training in the rehabilitation of elderly patients (60-75 years) following hip or knee arthroplasty.

DETAILED DESCRIPTION:
This randomized controlled trial will recruit 60 patients aged 60-75 years, within 3 months after total hip or knee arthroplasty, admitted to the Rehabilitation Unit of St. Jadwiga Hospital in Trzebnica. Participants will be randomly assigned to one of three groups: (i) body weight-supported treadmill group (n=20), (ii) antigravity treadmill group (n=20), or (iii) control group receiving conventional gait training (n=20). All patients will receive comprehensive daily therapy for 6 weeks, including kinesitherapy, ergotherapy, and physical therapy procedures under professional supervision.

ELIGIBILITY:
Inclusion Criteria:

* individuals who have recently undergone hip or knee joint arthroplasty surgeries aged 60 years and above.

Exclusion Criteria:

* cognitive impairments that prevent independent completion of research questionnaires
* history of consciousness disturbances, psychotic disorders, bipolar disorder, or other severe psychiatric illnesses
* functional status preventing independent ambulation (wheelchair-bound or bedridden patients; orthopedic devices such as crutches or walker allowed)
* refusal to participate in the study at any stage

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index | Baseline and after 6 weeks of intervention
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a 24-item questionnaire used to assess pain, stiffness, and physical function in patients with hip or knee osteoarthritis. Each item is scored on a scale from 0 to 4, with higher scores indicating greater severity. The total score is calculated as the sum of three subscales: pain (0-20 points), stiffness (0-8 points), and physical function (0-68 points), yielding a global score range of 0 to 96. Higher scores reflect worse joint function, greater pain, and more severe stiffness.

SECONDARY OUTCOMES:
Berg Balance Scale | Baseline and after 6 weeks of intervention
  The Berg Balance Scale (BBS) is a 14-item instrument assessing static and dynamic balance, scored 0 to 4 per item, with a total score ranging from 0 to 56. Higher scores indicate better balance and lower fall risk.
Patient Health Questionnaire | Baseline and after 6 weeks of intervention
  The Patient Health Questionnaire (PHQ-9) is a 9-item self-report scale measuring depressive symptoms, scored from 0 to 3 per item, with total scores ranging from 0 to 27. Higher scores indicate greater depression severity.
Perceived Stress Scale | Baseline and after 6 weeks of intervention
  The Perceived Stress Scale (PSS-10) is a 10-item instrument assessing perceived stress over the past month. Each item is rated 0-4, with total scores ranging from 0 to 40. Higher scores indicate higher perceived stress levels.
Falls Efficacy Scale-International | Baseline and after 6 weeks of intervention
  The Falls Efficacy Scale-International (FES-I) consists of 16 items assessing concern about falling during various activities. Items are scored from 1 to 4, with total scores ranging from 16 to 64. Higher scores reflect greater fear of falling.
Step Length | Baseline and after 6 weeks of intervention
  Step length (in centimetres) for the left and right lower limbs will be assessed during walking on an antigravity treadmill with integrated gait analysis. Values will be reported separately for each leg. An increase in step length is expected following the intervention.
Step Time | Baseline and after 6 weeks of intervention
  Step time (in milliseconds) for the left and right lower limbs will be measured during treadmill walking using an antigravity system. Values will be reported separately for each leg. A decrease in step time is expected following the intervention.
Stance Phase Duration | Baseline and after 6 weeks of intervention
  Stance phase duration (in percent of gait cycle) for the left and right lower limbs will be recorded during walking on an antigravity treadmill. Values will be reported separately for each leg.
Swing Phase Duration | Baseline and after 6 weeks of intervention
  Swing phase duration (in percent of gait cycle) for the left and right lower limbs will be assessed using gait analysis on an antigravity treadmill. Results will be reported separately for each leg.
Vertical Load | Baseline and after 6 weeks of intervention
  Vertical load (in percent of body weight) applied by the left and right lower limbs during stance will be measured using an antigravity treadmill with embedded load sensors. Values will be reported separately for each leg.

CONTACTS AND LOCATIONS:
Overall Officials: Justyna Mazurek, PhD, Principal Investigator — Wroclaw Medical University; Błażej Cieślik, PhD, Principal Investigator — Wroclaw University of Health and Sport Sciences; Joanna Szczepańska-Gieracha, Prof., Study Director — Wroclaw University of Health and Sport Sciences
Locations (1):
- St. Hedwig of Silesia Hospital in Trzebnica, Trzebnica, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No